CLINICAL TRIAL: NCT02651519
Title: Sleep Quality After Stellate-ganglion Block of Patients Undergoing Breast Cancer Operation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, associate proffessor, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015110302
Record Dates: First submitted 2016-01-05; First posted 2016-01-11 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2016-01

CONDITIONS: Sleep Deprivation
Keywords: bispectral index; regional cerebral oxygen saturation; Stellate-ganglion block
MeSH Terms: conditions — Sleep Deprivation | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): All patients undergoing breast cancer operation will be the treatment intervention with general anesthesia as an adjunct to stellate-ganglion block with saline.
  Interventions: Drug: saline
- stellate-ganglion block (Experimental): All patients undergoing breast cancer operation will be the treatment intervention with general anesthesia as an adjunct to stellate-ganglion block with 0.25% ropivacaine hydrochloride.
  Interventions: Drug: 0.25% ropivacaine hydrochloride

INTERVENTIONS:
Drug: 0.25% ropivacaine hydrochloride — stellate-ganglion block with 0.25% ropivacaine hydrochloride
  Arms: stellate-ganglion block
Drug: saline — stellate-ganglion block with saline
  Arms: Control

SUMMARY:
Stellate-ganglion block have been done safely for more than 60 years. It has proved to provide survivors of breast cancer with relief from hot flushes and sleep dysfunction with few or no side-effects. The aim of the present study is to evaluate postoperative sleep quality of patients undergoing breast cancer surgery with Stellate-ganglion block performed in the operation.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled (randomized, parallel group, concealed allocation), double-blinded trial. All patients undergoing breast cancer operation will be randomized 1:1 to the treatment intervention with general anesthesia as an adjunct to Stellate-ganglion block with 0.25% ropivacaine hydrochloride or saline. The objective of the trial is to evaluate the postoperative sleep quality of patients undergoing breast cancer operation with Stellate-ganglion block 0.25% ropivacaine hydrochloride or saline.

ELIGIBILITY:
Inclusion Criteria:

* At least18 years and pre-menopausal;
* scheduled to undergo elective breast cancer operation;
* American Society of Anaesthesiologists (ASA) risk classification I-II.

Exclusion Criteria:

* (1) patient refusal; (2) known hypersensitivity to the study medication (ropivacaine); (3) long-term use of opioids; (4) a history of psychiatric or neurological disease; (5) a preoperative Pittsburgh Sleep Quality Index (PSQI) global score higher than 6.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
sleep quality | first postoperative night
  The primary objective is to compare postoperative sleep quality, as measured using a bispectral index-Vista monitor during the first night after surgery.

SECONDARY OUTCOMES:
regional cerebral oxygen saturation | In the operation
  physiological parameter of regional cerebral oxygen saturation of all patients during the operation will be recorded.Regional cerebral oxygen saturation measured by near-infrared spectroscopy in the frontal lobe has been used previously to evaluate overall cerebral blood flow. The normal range of cerebral oxygen saturation is 55-80%.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-fei Tan, PhD,MD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jin F, Li XQ, Tan WF, Ma H, Fang B, Tian AY, Lu HW. Effects of ultrasound-guided stellate-ganglion block on sleep and regional cerebral oxygen saturation in patients undergoing breast cancer surgery: a randomized, controlled, double-blinded trial. J Clin Monit Comput. 2018 Oct;32(5):855-862. doi: 10.1007/s10877-017-0074-3. Epub 2017 Oct 17. PMID 29043600